CLINICAL TRIAL: NCT06125197
Title: A Phase I Open-Label, Dose-escalation Trial of Tumor Necrosis Factor Alpha and Interleukin-2 Coding Oncolytic Adenovirus (TILT-123) in Combination With Pembrolizumab in Patients With Immune Checkpoint Inhibitor Refractory Non-Small Cell Lung Cancer
Brief Title: Oncolytic Adenovirus TILT-123 With Pembrolizumab as Treatment for Refractory Non-Small Cell Lung Cancer
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: TILT Biotherapeutics Ltd. (Industry)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Tilt-T610; MK-3475-E46 (Other: Merck Sharp & Dohme LLC); KEYNOTE-E46 (Other: Merck Sharp & Dohme LLC)
Record Dates: First submitted 2023-10-31; First posted 2023-11-09 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms | interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- TILT-123 and Pembrolizumab (Experimental): Patients will receive multiple administrations of TILT-123 and Pembrolizumab.
  Escalation to the next dose of TILT-123 will occur when the safety data has been evaluated for patients in the preceding dose level.
  Interventions: Biological: TILT-123; Biological: KEYTRUDA®

INTERVENTIONS:
Biological: TILT-123 — Tumor necrosis factor alpha (TNFalpha) and Interleukin-2 (IL-2) coding oncolytic adenovirus TILT-123
  Other Names: Ad5/3-E2F-d24-hTNFa-IRES-hIL2 (TILT-123)
Biological: KEYTRUDA® — pembrolizumab, a monoclonal antibody binding PD-1
  Other Names: pembrolizumab; pembrolizumab (MK-3475)

SUMMARY:
This is an open label, Phase 1, dose escalation trial evaluating the safety of oncolytic adenovirus TILT-123 in combination with Pembrolizumab in patients with immune checkpoint inhibitor refractory non-small cell lung cancer.

ELIGIBILITY:
Inclusion Criteria:

Histologically confirmed NSCLC cancer which cannot be treated with curative intent with available therapies and is refractory to or progressing after anti-PD(L)1 immunotherapy or immunotherapies.

At least one tumor lesion (>15 mm or bigger) must be available for biopsy that in the opinion of the investigator, is accessible to repeated biopsies without major safety concerns.

The patient must have disease evaluable per RECIST 1.1

Have adequate organ function as defined in the following values below. Specimens must be collected within 10 days prior to the start of study treatment.

Hematological laboratory values

* Absolute neutrophil count (ANC): ≥1500/µL
* Platelets: ≥ 100 000/µL
* Hemoglobin: ≥9.0 g/dL or ≥5.6 mmol/L. Criteria must be met without packed red blood cell (pRBC) transfusion within the prior 2 weeks. Participants can be on stable dose of erythropoietin (≥ approximately 3 months.
* Leukocytes (WBC) > 3.0

Renal laboratory values

* GFR: >45 ml/min (Cockcroft-Gault formula).
* Hepatic laboratory values
* Total bilirubin: ≤1.5 ×ULN OR direct bilirubin ≤ULN for participants with total bilirubin levels >1.5 × ULN (excluding patients with Gilbert's disease)
* AST (SGOT) and ALT (SGPT): ≤2.5 × ULN (≤5 × ULN for participants with liver metastases)

Patients must be willing to use adequate forms of contraception from screening, during the trial, and for a minimum of 120 days after end of treatment.

ECOG/WHO performance score of 0-1 at screening.

Life expectancy longer than 3 months.

Exclusion Criteria:

* Has an active autoimmune disease that has required systemic treatment in past 2 years. Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency) and inhaled and topical treatments are not considered a form of systemic treatment and are allowed.

Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior the first dose of study drug.

Treated with any anti-cancer therapy within 30 days prior to the first virus injection.

Participants must have recovered from all AEs due to previous therapies to ≤Grade 1 or baseline. Participants with ≤Grade 2 neuropathy may be eligible.

Treated with a prior radiotherapy, including for palliative purposes, within 2 weeks of start of study treatment (before or after).

Treated with a prior therapy with an anti-PD-1, anti-PD-L1, or anti PD L2 agent or with an agent directed to another stimulatory or co-inhibitory T-cell receptor (e.g., CTLA-4, OX 40, CD137), and was discontinued from that treatment due to a Grade 3 or higher irAE.

History of myocarditis or congestive heart failure (as defined by New York Heart Association Functional Classification III or IV), cerebral stroke, unstable angina, serious uncontrolled cardiac arrhythmia, uncontrolled infection, or myocardial infarction 6 months prior to study entry.

History of myocardial infarction or cerebral stroke within the previous 12 months before screening or is not sufficiently recovered from an older infarction or cerebral stroke.

History of severe hepatic dysfunction.

History of Hepatitis B (defined as HBsAg reactive), Hepatitis C (defined as HCV RNA [qualitative] is detected) or HIV. No testing for Hepatitis B, Hepatitis C and HIV is required unless mandated by a local health authority.

History of coagulation disorder.

Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study, interfere with the participant's participation for the full duration of the study, or is not in the best interest of the participant to participate, in the opinion of the treating investigator.

Female patients who are pregnant, breastfeeding or intend to become pregnant. Women of child bearing potential who has a positive urine pregnancy test (within 72 hours) prior to treatment. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.

Has a known additional malignancy that is progressing or has required active treatment within the past 5 years. Participants with basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or carcinoma in situ (e.g., breast carcinoma, cervical cancer in situ) that have undergone potentially curative therapy are not excluded.

Has known active CNS metastases and/or carcinomatous meningitis.

Has an active infection requiring systemic therapy.

Has a history of (non-infectious) pneumonitis/interstitial lung disease that required steroids or has current pneumonitis/interstitial lung disease.

Has a known psychiatric or substance abuse disorder that would interfere with the participant's ability to cooperate with the requirements of the study.

Allergy to ingredients present in the investigational medicinal products (ingredients are listed in the protocol) ie. severe hypersensitivity (≥Grade 3) to pembrolizumab and/or any of its excipients.

Known contraindications to pembrolizumab.

Has had an allogenic tissue/solid organ transplant.

Has received a live or live-attenuated vaccine within 30 days prior to the first dose of study intervention. Administration of killed vaccines are allowed.

Has received radiation therapy to the lung that is >30Gy within 6 months of the first dose of trial treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Estimated)
Dates: Start 2024-07-23 (Actual); Primary Completion 2026-01-30 (Estimated); Study Completion 2026-05-30 (Estimated)

PRIMARY OUTCOMES:
Dose Escalation Phase | Day 1 to Day 85
  Incidence of DLT AEs in subjects with refractory NSCLC
Incidence of Adverse Events | Day 1 to Day 85
  Determine the safety and tolerability of the combination of TILT-123 and Pembrolizumab in patients with refractory non-small cell lung cancer by evaluating the number, frequency, and severity of adverse events using CTCAE v 5.0.

SECONDARY OUTCOMES:
Dose Escalation Phase MTD | Day 1 to Day 85
  Determine the Maximum Tolerated Dose in patients with refractory NSCLC

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Hoag Memorial Hospital Presbyterian, Newport Beach, California
  - UCLA Jonsson Comprehensive Cancer Center, Santa Monica, California